CLINICAL TRIAL: NCT00132704
Title: An Analysis of the Response of Human Tumor Microvascular Endothelium to Ionizing Radiation
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04-109
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Ovarian Neoplasms; Colorectal Neoplasms; Melanoma; Small Cell Lung Cancer; Liposarcoma
Keywords: Lung cancer metastases to the CNS (adenocarcinomas); Melanoma metastases to the CNS; Breast cancer metastases to the CNS (ductal carcinomas); Central nervous system gliomas; Colorectal cancers (adenocarcinomas); Ovarian cancers (papillary serous carcinomas); Endometrial cancers (endometrioid carcinomas); Cervical cancers (squamous cell carcinomas); Sarcomas (liposarcomas and leiomyosarcomas); Thoracic mesotheliomas; Colorectal cancers metastatic to the liver; Primary adenocarcinomas of the lung; Primary squamous cell carcinomas of the lung; Pancreatic Cancers-adenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Colorectal Neoplasms; Melanoma; Small Cell Lung Carcinoma; Liposarcoma; Adenocarcinoma; Carcinoma, Ductal; Endometrial Neoplasms; Carcinoma, Endometrioid; Uterine Cervical Neoplasms; Carcinoma, Squamous Cell; Sarcoma; Leiomyosarcoma | interventions — Radiation, Ionizing; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue

GROUPS / COHORTS (2):
- A: The experiments in Group A will be conducted in order to determine if human tumor microvascular endothelium displays similar dose parameters as mouse tumor endothelium, and if the microvascular endothelium of tumors of different types behaves in a similar fashion in its response to IR.
  Interventions: Radiation: Ionizing radiation (IR) therapy
- B: The experiments in Group B will be conducted in order to determine if tumor endothelium isolated to near homogeneity demonstrates dose parameters similar to those used in single dose radiotherapy of brain tumors.
  Interventions: Radiation: Ionizing radiation (IR)

INTERVENTIONS:
Radiation: Ionizing radiation (IR) therapy — Tumors will be sliced into 0.5cm fragments, incubated in culture medium and then irradiated to evaluate the kinetics and dose-dependencies of the endothelial apoptotic response. We will irradiate tumor fragments ex vivo at 0, 7, 13, 15, 17, and 25 Gy.
  Groups: A
Radiation: Ionizing radiation (IR) — Tissue fragments of a total quantity of at least a 4x4x4 cm3 will be required. For each tumor a paraffin block will also be made for routine staining and IHC. Endothelial cell populations (at least 500 cells) will then be exposed to radiation at 0, 7, 11, 13, 15, 17, and 25 Gy and harvested at 4, 5 and 8 hours post IR.
  Groups: B

SUMMARY:
Doctors will take some tissue from the tissue removed during surgery in order to study how the blood vessels of the tumor respond to radiation therapy. The tissue obtained will be used to determine how these tumor blood vessels respond to radiation therapy delivered to the tumor, after it has been removed. This radiation is delivered in the research lab. This research is being conducted in order to develop new methods to treat tumors by radiation therapy. No additional surgery will be performed to obtain these samples, and only materials that remain after all diagnostic testing has been completed will be used.

DETAILED DESCRIPTION:
The goal of this study is to determine if concepts established in mouse models of the tumor microvascular response to ionizing radiation (IR) therapy are applicable to human tumors in order to begin to establish that the engagement of the endothelial response is a valid target for IR in human tumors. A portion of tumor will be isolated from individuals who have signed informed consent for this protocol and are undergoing surgery on the Neurosurgery, Colorectal, and Gynecology, Head and Neck, Urology, and Hepatobiliary Services at Memorial Sloan-Kettering Cancer Center. Tumor tissue will be obtained from the surgical sample in pathology after adequate specimens have been obtained for diagnostic purposes. Tumor tissue will be irradiated ex vivo and the microvascular endothelial response will be determined. From specimens of adequate size, a pure tumor endothelial cell population will be isolated and the response to IR will be determined.

Primary Outcomes:

* To determine if human tumor microvascular endothelium displays similar dose parameters as mouse tumor endothelium.

Secondary Outcomes:

* To determine if tumor endothelium isolated to near homogeneity demonstrates dose parameters similar to those used in single dose radiotherapy of brain tumors.
* To determine if the microvascular endothelium of tumors of different types behaves in a similar fashion in its response to IR.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are felt to have adequate tumor volume for these studies, at least a 2 x 2 x 2 cm3 tumor by physical exam, imaging studies or colonoscopy reports
* Primary or recurrent tumors are eligible
* Patients must be suitable candidates for surgery
* Patients who have signed the informed consent

Exclusion Criteria:

* Patients who are not considered suitable candidates for surgery
* Patients who have received prior radiation therapy to the tumor being removed
* Patients who have received chemotherapy within 6 months of tumor removal
* Patients who are pregnant
* Patients may choose to be excluded at any time
* Minors are excluded from this study because there are expected to be very few minors with the tumor types which the investigators are evaluating in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: undergoing surgery on the Neurosurgery, Hepatobiliary, Colorectal, Urology, Head and Neck, Gynecology, GMT and Thoracic Services at Memorial Sloan- Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2004-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
apoptotic response | 2 years
  The peak apoptotic radiation response will be obtained for each of the tumor type and the result compared to that of the mouse experiments in Garcia-Barros (no formal testing only qualitative statements).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: (Memorial Sloan-Kettering Cancer Center) — http://mskcc.org